CLINICAL TRIAL: NCT01538498
Title: A Clinical Trial to Develop a Peritoneal Carcinomatosis Index (PCI) in Ovarian
Brief Title: Development for the Peritoneal Carcinomatosis Index (PCI) in Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Sang-Yoon Park, Chief, Center for Uterine Cancer, National Cancer Center, Korea
Other Study IDs: NCCCTS-08-309
Record Dates: First submitted 2012-02-17; First posted 2012-02-24 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Ovarian Cancer
Keywords: PCI; Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
* Primary objectives: To develop peritoneal carcinomatosis index (PCI) for ovarian cancer, tubal cancer and primary peritoneal cancer that can represent perioperative intraperitoneal tumor burden objectively
* Secondary objectives: To establish the relationship and find out clinical significance between PCI, tumor location and tumor characteristics

DETAILED DESCRIPTION:
Patients with primary ovarian cancer

* Informed consent
* Digital photography & Checking PCI (tumor size, number, and Characteristics)
* Postoperative surveillance(tumor marker, image and physical examination)

  1. Developing the best fitting PCI model to reflect recurrence-free survival and overall survival

     * Selection of items
     * Weighting by items and tumor characteristics
  2. Analysis of prognostic impact of PCI compared to conventional staging system (FIGO stage) for ovarian cancer

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative clinical diagnosis of ovarian cancer, tubal cancer, and primary peritoneal carcinoma (all stage)
2. Available preoperative image study (CT and/or MRI and/or PET)
3. Patients who gave a written informed consent
4. Patients must be surgical candidate considering medical and psychological condition

Exclusion Criteria:

* Patients who refuse to participate or want to withdraw at anytime.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * primary ovarian cancer
  * non-neoadjuvant
  * Debulking operation
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2008-04; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Devleopment for the peritoneal carcinomatosis index (PCI) | 55 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea